CLINICAL TRIAL: NCT03198104
Title: Assessing Kids for Liver Inflammation and Fibrosis Using Non-invasive MRI
Acronym: Kids4LIFe
Status: Completed | Type: Observational
Sponsor: Perspectum (Industry)
Collaborators: Children's Memorial Health Institute, Poland (Other)
Responsible Party: Sponsor
Other Study IDs: PJM076
Record Dates: First submitted 2017-06-19; First posted 2017-06-23 (Actual); Last update posted 2019-08-30 (Actual); Status verified 2019-08

CONDITIONS: Non-alcoholic Steatohepatitis; Liver Diseases; Liver Fibroses; Autoimmune Hepatitis; Liver Cirrhoses
Keywords: Multiparametric MR Imaging; Paediatric
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Liver Diseases; Liver Cirrhosis; Hepatitis, Autoimmune

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Liver biopsy and histology.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Liver disease: Paediatric patients (50-60 pts.) with liver disease who are scheduled for an ultrasound-guided liver biopsy as part of their standard care - these patients will be scanned using MRI and fibroscan, then will proceed through standard care pathway to receive blood tests and a liver biopsy. Findings from the fibroscan, blood tests and liver biopsy will be compared to the MRI data to determine it's accuracy in detecting and distinguishing different types of liver disease.
  Interventions: Device: MRI
- Autoimmune Hepatitis Group (AIH): Paediatric patients who have been diagnosed with autoimmune hepatitis and are about to initiate pharmacological treatment (15-30 pts.) will be scanned using MRI and fibroscan, then proceed through the standard care pathway to receive repeated blood tests and liver biopsies throughout treatment. MRI and fibroscan will be repeated before each liver biopsy. Findings from the fibroscan, blood tests and liver biopsy will be compared to MRI data to determine it's accuracy in monitoring liver disease.
  Interventions: Device: MRI
- Healthy Volunteers: Healthy volunteers (20-30 children) will be scanned using MRI and fibroscan and used as healthy controls.
  Interventions: Device: MRI

INTERVENTIONS:
Device: MRI
  Other Names: LiverMultiScan

SUMMARY:
This is a prospective observational study which will recruit up to 100 paediatric participants over a period of 30 months to determine whether MRI is as accurate at detecting, distinguishing, and monitoring liver disease as current standard of care techniques such as liver biopsy and fibroscan.

DETAILED DESCRIPTION:
The most serious pandemic facing Europe is fatty liver disease and non-alcoholic steatohepatitis (NASH). The main causal factor is obesity: according to recent statistics 11.8m-16.3m European children are overweight, of which 2.9m - 4.4m are obese. Unfortunately, current techniques for the diagnosis and monitoring of liver disease in children are poor. Available methods are either insensitive, such as blood tests, or invasive, i.e. liver biopsy, which is risky, painful, and costly. Although it is currently considered to be the gold standard for tissue assessment, liver biopsy has severe limitations, one of which is that it samples only a tiny fraction of the liver, and so it cannot give a representative diagnosis when liver disease is regional. Early determination of liver diseases in children, could have a significant impact on changing the course of illness and on the proper treatment management.

Perspectum Diagnostics have demonstrated that multiparametric MR imaging can, for the first time, allow accurate, non-invasive detection of liver fibrosis/inflammation in adults, and predict clinical outcomes (1,2). However, liver disease in children differs from adults in aetiology, natural history and pathological findings (3,4).

This study will investigate whether non-invasive multiparametric MR imaging of the liver can accurately and reproducibly detect, distinguish and track progression of different forms of liver disease in the paediatric population. To achieve this, children with liver disease who are scheduled to undergo liver biopsy and blood tests as part of their standard care will be recruited. Non-invasive, pain-free MRI scanning will be used to measure fibrosis, iron content and fat content of liver tissue and compare these results to the findings of the liver biopsy that is being performed as standard care. Children who are scheduled to receive repeated liver biopsies to monitor their response to the treatment of autoimmune hepatitis as part of their usual care will also be included. Repeated MRI scans will be performed and compared with the results of biopsy findings.

ELIGIBILITY:
Inclusion Criteria:

Group 1 (Liver disease):

* Male or female between 6 - 18 years of age
* Male or female aged between 1-10 years of age and scheduled to receive an MRI under anesthesia as part of their standard care.
* Scheduled to receive an ultra-sound guided liver biopsy as part of their usual care
* Participant and guardian are willing and able to give assent and consent for participation in the study

Group 2 (AIH):

* Male or female between 6 - 18 years of age
* Male or female aged between 1-10 years of age and scheduled to receive an MRI under anesthesia as part of their standard care.
* Diagnosed with autoimmune hepatitis and due to begin liver-biopsy monitored treatment as part of their usual care
* Participant and guardian are willing and able to give assent and consent for participation in the study

Group 3 (Healthy controls):

* Male or female between 6 - 18 years of age (age-matched with Group 1)
* Lean, defined as within interquartile range for age and sex-matched childhood BMI growth charts
* Healthy, with no active medical condition requiring treatment, including diabetes, hypertension, psoriasis and any chronic gastrointestinal disorder
* Participant and guardian are willing and able to give assent and consent for participation in the study

Exclusion Criteria:

* The participant may not enter the study if they have any contraindication to magnetic resonance imaging (inc pregnancy, extensive tattoos, pacemaker, shrapnel injury, severe claustrophobia).
* Any other cause, including a significant disease or disorder which, in the opinion of the investigator, may either put the participant at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Participants aged between 6-18 years of age with liver disease who are scheduled to receive a liver biopsy as part of their usual care and age-matched healthy volunteers aged 6-18 years of age. Participants between 1-10 years of age who are scheduled to receive an MRI scan under anesthesia as part of their standard care will also be recruited.
Sampling Method: Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Multiparametric non-invasive MRI of liver tissue in detecting and distinguishing different forms of paediatric liver disease. | 30 months
  Measurements using multiparametric MRI and comparison of these results with liver biopsy findings.

SECONDARY OUTCOMES:
Determining use of MRI in measuring changes in liver disease within patient. | 30 months
  Measurements using repeated MRI and comparison of these results with repeated paediatric liver biopsy findings throughout the course of treatment for autoimmune hepatitis.

CONTACTS AND LOCATIONS:
Overall Officials: Rajashi Banerjee, MD, PhD, Study Director — Perspectum Diagnostics; Piotr Socha, MD, Principal Investigator — Children's Memorial Health Institute, Poland
Locations (1):
- Children's Memorial Health Institute Poland, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No
All data stored from patients (including MRI data files) will be anonymised during upload to the custom-built data management system that is being designed specifically for this study. No project partner will be able to access identifiable information (with the exception of the medical team who will upload the data).

REFERENCES:
- [Derived] Janowski K, Shumbayawonda E, Dennis A, Kelly M, Bachtiar V, DeBrota D, Langford C, Thomaides-Brears H, Pronicki M, Grajkowska W, Wozniak M, Pawliszak P, Chelstowska S, Jurkiewicz E, Banerjee R, Socha P. Multiparametric MRI as a Noninvasive Monitoring Tool for Children With Autoimmune Hepatitis. J Pediatr Gastroenterol Nutr. 2021 Jan 1;72(1):108-114. doi: 10.1097/MPG.0000000000002930. PMID 32925554